CLINICAL TRIAL: NCT06505564
Title: VR-based Avatar Therapy for Treatment of Auditory Hallucinations in Patients With Schizophrenia 2023-SUD-3446
Brief Title: VR-based Avatar Therapy for Treatment of Auditory Hallucinations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Collaborators: University of Barcelona (Other); Parc Sanitari Sant Joan de Déu (Other); Fundació Sant Joan de Déu (Other); Uniwersytet Medyczny w Łodzi (Unknown)
Responsible Party: Principal Investigator, Gábor Csukly, Associate professor, Semmelweis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VR-AT-SCH 2023-SUD-3446
Record Dates: First submitted 2024-07-02; First posted 2024-07-17 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Hallucinations, Auditory; Schizophrenia Spectrum and Other Psychotic Disorders
Keywords: Virtual reality; AVATAR therapy; Auditory verbal hallucation; Schizophrenia spectrum disorder
MeSH Terms: conditions — Hallucinations; Schizophrenia Spectrum and Other Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: This study aims to evaluate the efficacy of AVATAR therapy in patients with schizophrenia spectrum disorder using a single-group pre-post design with a waiting list control period. Initially, all patients will undergo a 12-week waiting list control period without treatment. Following this phase, participants will receive AVATAR therapy consisting of 7 sessions over 12 weeks. Comprehensive assessments will be conducted before and at the end of the waiting list period, with post-therapy assessments following the intervention. Evaluations by caregivers and therapists will also be included to provide comprehensive insights into the therapy's effectiveness and overall impact.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AVATAR therapy (Experimental): All participants will initially undergo a 12-week waiting period (control period) starting from the initial screening at week 0. Baseline assessments will be conducted at week 12. Subsequently, participants will receive AVATAR therapy for 12 weeks. Post-therapy assessments will be conducted at week 24. Caregivers and therapists will also provide evaluations to gather additional insights into the therapy's impact
  Interventions: Behavioral: AVATAR therapy

INTERVENTIONS:
Behavioral: AVATAR therapy — In the initial phase of treatment, patients collaborate with therapists to visualize the source of their auditory hallucinations. Therapists adjust their voice to match the hallucinations, prompting patients to recall key statements for future sessions. Subsequent sessions involve dialogues with a computerized avatar. Using the altered voice, therapists interact in real-time through the avatar, engaging patients in role-playing. They alternate between the avatar and supportive therapist roles to empower patients with positive affirmations and discussions. Sessions last approximately 50 minutes, utilizing Oculus Rift VR headsets and noise-cancelling headphones to enhance immersion. HEKA VR software adjusts avatar proximity, and patients have the option to record dialogues for home use and sharing. Therapists receive bi-weekly supervision from HEKA VR-trained colleagues. Participants continue their regular medication prescribed by their psychiatrists alongside this experimental therapy

SUMMARY:
The primary aim of this study is to evaluate the safety and efficacy of AVATAR therapy, developed to address residual auditory hallucinations persisting despite medication in schizophrenia spectrum disorder. The intervention aims to reduce the intensity and frequency of these symptoms, as well as alleviate associated depressive and anxiety symptoms, using a virtual reality (VR)-assisted intervention developed for this purpose by the Danish company HEKA VR. The study will be a pre-post non-invasive, waiting list-controlled study, enrolling 30 patients from three clinical sites (Hungary, Spain, Poland).

The study centers around administering therapy based on VR over a 12-week period, comprising a total of 7 sessions. These sessions are conducted individually and last 50 minutes each. The psychotherapist leading the sessions adheres to a strict protocol defined by the method's developers.

During the intervention, VR technology is used to simulate the source of distressing auditory hallucinations. The therapist facilitates coping with these experiences externalized in this way through simulated conversations, supporting the development of more adaptive responses.

Patients undergo a comprehensive cross-sectional evaluation of their condition before and after the intervention, including assessments of symptom severity, quality of life, and their experience with the method. The intervention is conducted with constant monitoring for possible adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia spectrum disorder according to DSM-5,
* Age 18 or older,
* The fluent use of the spoken language at the site (Hungarian/Spanish/Polish),
* Informed consent provided by the patient or their caregiver after being informed about the research procedure
* Stable medication dosage for at least 4 weeks prior to recruitment,
* Regular psychiatric follow-up,
* Experience of auditory hallucinations for at least three months (PANSS hallucination score of at least 3 points),
* Meeting the remission criteria described by Andreasen, except for the score related to auditory hallucinations

Exclusion Criteria:

* Inability to identify a single dominant voice that is the subject of the intervention,
* Lack of cooperation,
* Intellectual disability based on medical history,
* Regular substance abuse
* Central nervous system injury or neurological disease that affects cognitive performance,
* Suicidal risk
* Aversion to virtual reality,
* Severe visual impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in symptom severity | Week 0, Week 12, Week 24
  Positive and Negative Syndrome Scale: Assesses overall symptom severity in schizophrenia spectrum disorders, including positive symptoms (e.g., hallucinations, delusions), negative symptoms (e.g., affective flattening, social withdrawal), and general psychopathology (e.g., anxiety, depression).The scale is administered through a semi-structured interview by trained clinicians. The minimum possible score for positive and negative symptoms is 7 points, and the maximum possible score is 49 points. For general symptomatology, the possible minimum score is 16 points, and the maximum score is 112 points. The overall score can range from 30-210. Higher scores indicate greater symptom severity.
Change in severity of auditory hallucinations | Week 0, Week 12, Week 24
  Psychotic Symptom Rating Scales: Evaluates the severity of auditory hallucinations and associated delusions, including frequency, duration, loudness, and disruption. The scale is administered through a semi-structured interview by trained clinicians. The scale comprises 17 items of the mentioned specific dimensions of hallucinations and delusions, with each item being rated from 0 (absent) to 4 (severe). The total score range for the test is 0 to 68, where lower scores indicate reduced severity of hallucinatory experiences.
Change in beliefs about voices in schizophrenia spectrum disorder | Week 0, Week 12, Week 24
  Beliefs About Voices Questionnaire-Revised: A self-report questionnaire designed to assess individuals' beliefs about auditory hallucinations (e.g.: how important the voices are to the individual, perceived control, emotional reactions elicited by the voices. The scale comprises 35 items, with each item being rated from 0 to 3. The total score range for the test is 0-105, where lower scores indicate reduced distress and improved coping with hallucinatory experiences.

SECONDARY OUTCOMES:
Change in comorbidity (depression) | Week 0, Week 12, Week 24
  Calgary Depression Scale for Schizophrenia: Evaluates the severity of depressive symptoms in patients with schizophrenia. It is administered through a semi-structured interview, conducted by trained clinicians. The scale comprises 9 items, with each item being rated from 0 (absent) to 3 (severe). The total score range for the test is 0 to 27, where lower scores indicate reduced depressive symptoms and improved comorbidity management.
Change in comorbidity (anxiety) | Week 0, Week 12, Week 24
  State-Trait Anxiety Inventory: A self-report questionnaire designed to assess anxiety levels in individuals. It distinguishes between two types of anxiety:
  State Anxiety: Refers to temporary feelings of anxiety that are situational and can fluctuate based on current circumstances.
  Trait Anxiety: Refers to a stable characteristic of an individual, reflecting a general tendency to respond with anxiety across various situations.
  The test consists of 40 items, with 20 items dedicated to measuring state anxiety and 20 items for trait anxiety. Respondents indicate how they feel on a scale from 1 (not at all) to 4 (very much so). Scores for each sub-scale can range from 20 to 80, with higher scores indicating greater levels of anxiety.
Change in health-related quailty of life | Week 0, Week 12, Week 24
  EuroQol 5-Dimension 5-Level Scale: A standardised instrument for measuring health-related quality of life. It consists of two main components: the descriptive system and the visual analog scale.
  The descriptive system includes five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Respondents rate their health status in each dimension on a scale from 1 (no problems) to 5 (extreme problems), resulting in a profile that can be converted into a single index value.
  The visual analog scale allows individuals to rate their overall health on a scale from 0 (worst imaginable health) to 100 (best imaginable health).
Change in subjective well-being | Week 0, Week 12, Week 24
  World Health Organisation Well-being Index: A brief self-report measure designed to assess subjective well-being and overall quality of life. Comprising five items, the index evaluates key aspects of emotional well-being over the past two weeks, including mood, energy, and general happiness. Respondents rate each item on a scale from 0 (at no time) to 5 (all of the time), resulting in a total score ranging from 0 to 25. Higher scores indicate better well-being and psychological health.
Change in emotion regulation | Week 0, Week 12, Week 24
  Emotion Regulation Questionnaire: A self-report measure designed to assess individual differences in the habitual use of two emotion regulation strategies: cognitive reappraisal and expressive suppression. The questionnaire consists of 10 items, with respondents indicating their agreement on a scale from 1 (strongly disagree) to 7 (strongly agree). The possible total scores range from 10 to 70, with higher scores on cognitive reappraisal typically associated with better psychological outcomes, while higher scores on expressive suppression may be linked to various negative effects.
Change in self-efficacy | Week 0, Week 12, Week 24
  General Self-Efficacy Scale: A self-report scale designed to assess perceived self-efficacy in coping with various stressors and challenges. The scale consists of 10 items that assess confidence in one's ability to handle different situations and overcome obstacles. Respondents rate each item on a scale from 1 (not at all true) to 4 (exactly true). Scores can range from 10-40, with higher scores indicate greater perceived self-efficacy.

OTHER OUTCOMES:
Patient satisfaction | Week 24
  Patient Satisfaction Questionnaire: The questionnaire evaluates overall satisfaction with AVATAR therapy sessions by using open-ended questions and Likert scales. This questionnaire was created by the research team and adjusted specifically for this therapy.
Therapist opinion | Week 24
  Therapist Opinion Questionnaire: The questionnaire assesses therapists' subjective opinions on the effectiveness and feasibility of AVATAR therapy by using open-ended questions and Likert scales. This questionnaire was created by the research team and adjusted specifically for this therapy.
Caregiver opinion | Week 24
  Caregiver Opinion questionnaire: The questionnaire measures caregivers' perspectives on the impact of AVATAR therapy on patient well-being and daily functioning by using a questionnaire that includes open-ended questions and Likert scales. his questionnaire was created by the research team and adjusted specifically for this therapy.
Side effects | After every therapy session between Week 13 and Week 23
  Simulator sickness questionnaire: A self-report tool used to assess symptoms of simulator sickness, which can occur during virtual reality. The questionnaire consists of 16 items that measure various symptoms associated with simulator sickness, including nausea, disorientation, and eye strain. Respondents rate the severity of each symptom on a scale from 0 (none) to 3 (severe). The total score ranges from 0-48, with higher scores indicating greater severity of simulator sickness.
Cost-effectiveness analysis of the intervention | Week 0, Week 12, Week 24
  Conduct a thorough cost-effectiveness analysis within health economics, assessing the economic impact of the healthcare intervention under investigation through meticulous collection and analysis of healthcare utilization data, intervention-related costs, and health outcomes data. This will be achieved using a detailed demographic questionnaire, which includes information on disease duration (time since diagnosis), illness progression (such as frequency and duration of hospital stays), direct and indirect costs of care (such as medication costs, productivity loss, travel expenses, and caregiver burden), and patient living conditions (covering socio-economic status, employment, and living arrangements). The health economic evaluation will involve repeated administration of this questionnaire, ensuring adherence to established best practices and ethical standards

CONTACTS AND LOCATIONS:
Locations (4):
- Semmelweis University, Budapest, Hungary
- Uniwersytet Medyczny w Łodzi, Lodz, Poland
- Spain (2):
  - Unitat de Recerca del Parc Sanitari Sant Joan de Déu, Barcelona
  - University of Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: No